CLINICAL TRIAL: NCT06096753
Title: Comparative Evaluation of Gnathological Function With Bruxoff® in Edentulous Patients With Immediate Load Full-arch Restorations (Columbus Bridge ProtocolTM) vs Toothed Patients: a Pilot Study
Brief Title: Comparative Evaluation of Gnathological Function With Bruxoff®
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Turin, Italy (Other)
Collaborators: Prof. Andrea Deregibus (Unknown); Dr. Armando Crupi (Unknown); Dra. Giulia Ambrogio (Unknown); Dr. Andrea Roccuzzo (Unknown); Miss Lisa Sannicolo (Unknown)
Responsible Party: Principal Investigator, Francesco Pera, prof., University of Turin, Italy
Other Study IDs: Bruxoff
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Gnathological Function
Keywords: Bruxism; Immediate-load implants; Columbus Bridge Protocol; Bruxoff; Gnathological function
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: The Test Group will include patients rehabilitated according to the full-arch method (Columbus Bridge ProtocolTM) with immediate loading for at least 6 months prior to the first nocturnal recording using Bruxoff®.
  Interventions: Device: Bruxoff gnathological function analysis
- Control Group: The Control Group will include healthy subjects and volunteers awaiting implant-prosthetic rehabilitation of intercalated edentulism (i.e. single-tooth gap) who have natural dentition up to the first molar.
  Interventions: Device: Bruxoff gnathological function analysis

INTERVENTIONS:
Device: Bruxoff gnathological function analysis — The recordings will be carried out for 3 randomly selected nights within 3 weeks, with at least 4 hours of sleep per night.

SUMMARY:
This study aims to compare the gnathological function of edentulous patient rehabilitated according to the full-arch method (Columbus Bridge Protocol™) with immediate loading with that of dentate patients, through at-home night-time monitoring with Bruxoff® device.

DETAILED DESCRIPTION:
Dental implants are now widely used in dentistry for the rehabilitation of partially or totally edentulous arches. These devices have shown excellent clinical success and are considered a reliable long-term treatment(1). In particular, the rehabilitation of the complete arch with immediate loading supported by maxillary implants has now become a safe and reliable procedure capable of rehabilitating the patient with residual or totally edentulous teeth. A fixed prosthesis supported by implants performed according to an immediate loading protocol represents a valid therapeutic option for the rehabilitation of totally edentulous patients, both from the point of view of patient satisfaction and masticatory performance(2,3,4).

Among the various protocols available in the literature, the one called Columbus Bridge Protocol™, developed by the prosthetic school of the University of Genoa, consists in the rehabilitation of one or both jaws with the insertion of a variable number of 4 to 6 dental implants followed by immediate loading(5). This rehabilitation has been documented to be a reliable implant-prosthetic solution in terms of survival and implant success in the medium and long term(2,6). However, considering the current scientific evidence, there is a lack of information relating to possible alterations in muscle activity following this implant-prosthetic rehabilitation.

For the evaluation of EMG activity of the stomatognathic system, the School of Turin has, for a decade now, tested and validated the use of Bruxoff® portable device for the evaluation of nocturnal bruxism, demonstrating a sensitivity and specificity of 91.6 % and 84.6% respectively (7,8).

Bruxoff® is a portable holter that uses 3 recording channels: 2 for recording the surface electromyographic signals (sEMG) of the two masseter muscles with concentric electrodes positioned on the two muscles (CoDe®: Concentric Detection, Spes Medica, Battipaglia, Italy), and one for heart rate detection (ECG) with a strap incorporating three surface electrodes positioned on the left side of the chest (7,13).

Patients who have been rehabilitated with a full-arch for at least 6 months at the Dental School of Turin and subjects waiting for implant-prosthetic rehabilitation of intercalated edentulism (i.e. single-tooth gap) will be involved.

The recordings will be carried out for 3 randomly selected nights within 3 weeks, with at least 4 hours of sleep per night, according to the method evaluated by Deregibus et al. In particular, the subjects will be instructed to perform 3 maximum voluntary contractions (Maximum Voluntary Clenching, MVC) lasting 2 seconds each and spaced by 5 seconds of rest at the beginning of the recording. The highest measurement among the MVCs is used to normalize the EMG values as a percentage of MVCs. The processing of the data will be carried out automatically and standardized using Bruxmeter software (Bruxmeter®, Spes Medica, Battipaglia, Italy) capable of processing the data recorded from the masseter muscles (surface electromyographic signal) and from the heart (cardiotachymetric signal).

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Age >18 years
* M/F sex
* Good general state of health
* Absence of clinical symptoms of bruxism, i.e. sore masticatory muscles(10,11)
* Good level of oral hygiene (assessed with FMPS <25%)
* FMBS <25%

Exclusion Criteria (9):

* Age <18 years
* Presence of severe psychiatric pathologies
* Presence of neuromuscular diseases/ severe neurodegenerative diseases
* Presence of diabetes or other metabolic diseases
* Pharmacological treatment with drugs that compromise the neuromuscular system
* Pharmacological treatment with antipsychotic drugs
* Presence of severe chronic diseases
* Cognitive disability
* Acute inflammation
* Presence of an oncological condition
* Smoking (>10 cigarettes per day) Individuals with alcohol or drug addiction will be excluded. Subjects will also be asked not to consume caffeine, alcohol and tobacco in the 6 hours before starting the night recording with Bruxoff®(12).

Patients with implants affected by peri-implant pathology will be excluded from the Test Group.(15) Subjects suffering from periodontal disease (Stage III/IV Grade B/C) will be excluded from the Control Group (16).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The subjects to be included in the study will be chosen from the list of patients rehabilitated according to the immediate-loading full-arch method (Columbus Bridge Protocol™) at the SCDU of Oral Rehabilitation, Maxillofacial Prosthetics and Dental Implantology (University of Turin) (Test Group) and from the list of subjects waiting for implant-prosthetic rehabilitation of intercalated edentulism (i.e. single-tooth implant) (Control Group).
  The subjects of the Control Group will be matched with a 1:1 ratio for the variables sex and age (±5 years) to the patients of the Test Group.
  Given the nature of the study (i.e. pilot study), the calculation of the sample size was not possible in the planning phase of the study. However, based on the evidence obtained from similar studies(7), 10 subjects per group are considered sufficient to test this method.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Masseter contractions | Night 1, Night 2, Night 3
  Number and type of masseter contractions (tonic/phasic/mixed)
Bruxism episodes | Night 1, Night 2, Night 3
  Number of possible episodes of nocturnal bruxism in total and per hour of sleep
Heart rate | Night 1, Night 2, Night 3
  Average heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pera, Prof., Principal Investigator — University of Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howe MS, Keys W, Richards D. Long-term (10-year) dental implant survival: A systematic review and sensitivity meta-analysis. J Dent. 2019 May;84:9-21. doi: 10.1016/j.jdent.2019.03.008. Epub 2019 Mar 20. PMID 30904559
- [Background] Pera P, Menini M, Pesce P, Bevilacqua M, Pera F, Tealdo T. Immediate Versus Delayed Loading of Dental Implants Supporting Fixed Full-Arch Maxillary Prostheses: A 10-year Follow-up Report. Int J Prosthodont. 2019 Jan/Feb;32(1):27-31. doi: 10.11607/ijp.5804. PMID 30677109
- [Background] Dellepiane E, Pera F, Zunino P, Mugno MG, Pesce P, Menini M. Oral Health-Related Quality of Life and Full-Arch Immediate Loading Rehabilitation: An Evaluation of Preoperative, Intermediate, and Posttreatment Assessments of Patients Using a Modification of the OHIP Questionnaire. J Oral Implantol. 2020 Dec 1;46(6):540-549. doi: 10.1563/aaid-joi-D-19-00274. PMID 33494102
- [Background] Pesce P, Menini M, Furnari M, Pera F, Tealdo T, Pera P. Gastric and masticatory performances in full-arch immediate loading rehabilitated patients. J Oral Rehabil. 2015 Sep;42(9):663-9. doi: 10.1111/joor.12301. Epub 2015 Apr 16. PMID 25882620
- [Background] Tealdo T, Bevilacqua M, Menini M, Pera F, Ravera G, Drago C, Pera P. Immediate versus delayed loading of dental implants in edentulous maxillae: a 36-month prospective study. Int J Prosthodont. 2011 Jul-Aug;24(4):294-302. PMID 21716965
- [Background] Deregibus A, Castroflorio T, Bargellini A, Debernardi C. Reliability of a portable device for the detection of sleep bruxism. Clin Oral Investig. 2014 Nov;18(8):2037-43. doi: 10.1007/s00784-013-1168-z. Epub 2013 Dec 28. PMID 24374575
- [Background] Castroflorio T, Deregibus A, Bargellini A, Debernardi C, Manfredini D. Detection of sleep bruxism: comparison between an electromyographic and electrocardiographic portable holter and polysomnography. J Oral Rehabil. 2014 Mar;41(3):163-9. doi: 10.1111/joor.12131. Epub 2014 Jan 7. PMID 24417585
- [Background] Saczuk K, Lapinska B, Wilmont P, Pawlak L, Lukomska-Szymanska M. The Bruxoff Device as a Screening Method for Sleep Bruxism in Dental Practice. J Clin Med. 2019 Jun 28;8(7):930. doi: 10.3390/jcm8070930. PMID 31261634
- [Background] Shimada A, Castrillon EE, Svensson P. Revisited relationships between probable sleep bruxism and clinical muscle symptoms. J Dent. 2019 Mar;82:85-90. doi: 10.1016/j.jdent.2019.01.013. Epub 2019 Feb 1. PMID 30716450
- [Background] Lobbezoo F, Ahlberg J, Raphael KG, Wetselaar P, Glaros AG, Kato T, Santiago V, Winocur E, De Laat A, De Leeuw R, Koyano K, Lavigne GJ, Svensson P, Manfredini D. International consensus on the assessment of bruxism: Report of a work in progress. J Oral Rehabil. 2018 Nov;45(11):837-844. doi: 10.1111/joor.12663. Epub 2018 Jun 21. PMID 29926505
- [Background] Bertazzo-Silveira E, Kruger CM, Porto De Toledo I, Porporatti AL, Dick B, Flores-Mir C, De Luca Canto G. Association between sleep bruxism and alcohol, caffeine, tobacco, and drug abuse: A systematic review. J Am Dent Assoc. 2016 Nov;147(11):859-866.e4. doi: 10.1016/j.adaj.2016.06.014. Epub 2016 Aug 10. PMID 27522154
- [Background] Mizumori T, Sumiya M, Kobayashi Y, Inano S, Yatani H. Prediction of sleep bruxism events by increased heart rate. Int J Prosthodont. 2013 May-Jun;26(3):239-43. doi: 10.11607/ijp.3305. PMID 23626977
- [Background] Farina D, Cescon C. Concentric-ring electrode systems for noninvasive detection of single motor unit activity. IEEE Trans Biomed Eng. 2001 Nov;48(11):1326-34. doi: 10.1109/10.959328. PMID 11686631
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952